CLINICAL TRIAL: NCT03341546
Title: Validation of a Computational Model to Estimate Patient Anterior-posterior Dimension From an Abdominal Radiograph
Brief Title: Estimating Patient Size From a Single Radiograph
Acronym: VocMepAdar
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Mark Worrall, Radiation Protection Adviser, NHS Tayside
Other Study IDs: 2017RA01
Record Dates: First submitted 2017-10-31; First posted 2017-11-14 (Actual); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Testing a Computational Model to Estimate Patient Size

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: 20 patients referred to Ninewells Hospital radiology department for an anterior-posterior abdomen x-ray examination. All of these patients will have a measurement of their anterior-posterior depth before undergoing their x-ray examination. An estimate of their anterior-posterior depth will then be made from their x-ray image using the computational model.
  Interventions: Other: A single measurement of the patient's abdominal depth

INTERVENTIONS:
Other: A single measurement of the patient's abdominal depth — A single measurement of the patient's anterior-posterior abdominal depth

SUMMARY:
A computational model has been created to estimate the abdominal depth of a patient from a single x-ray image. The model has been tested using phantoms and found to be accurate; this study aims to test the accuracy of the model with patients and in a clinical setting.

This will be achieved by enrolling patient's who have already been referred for an anterior-posterior abdomen x-ray examination to the trial, taking a physical measurement of their anterior-posterior abdominal depth and then comparing this measured value with a value as estimated using the computational model based on the patient's x-ray image.

DETAILED DESCRIPTION:
A non-commercial computational model has been developed in-house to estimate the patient's anterior-posterior or lateral depth using the radiographic image and the known exposure factors with which it was undertaken. This model has been tested using single composition phantoms and found to be accurate. If it was found to be accurate for real clinical examinations, this would automate the measurement of patient size and give institutions the estimate of patient size required for local paediatric patient dose audit. In turn, this would provide the national data required to propose national reference values for paediatric x-ray examinations, which would give all institutions an important comparator for their performance. This would lead to optimisation in those sites most requiring it; nationally, paediatric x-ray imaging would improve in time.

This pilot study is necessary to determine if the computational model is accurate enough to be relied upon. Accuracy will be determined by comparing the estimate made by the computational model for each patient with an actual measurement of the patient's anterior-posterior abdomen depth made at the time of the examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Referred to Ninewells Hospital for an anterior-posterior abdomen x-ray examination

Exclusion Criteria:

* Patients unable to give consent
* Patients who have had a contrast injection in the previous 24 hours
* Patients suffering abdominal pain at the time of the examination

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory outpatients attending Ninewells Hospital's radiology department for an anterior-posterior abdomen x-ray examination
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Vinnicombe, MD, Study Chair — University of Dundee
Locations (1):
- NHS Tayside, Dundee, Angus, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Cohort
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient Cohort
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of the Computational Model
Description: The computational model was used to estimate the patient's anterior-posterior abdominal depth using the digital radiographic image, the exposure factors with which it was acquired and a priori knowledge relating to the x-ray unit and digital detector.
  The outcome measure was the accuracy with which the computational model estimates the patient's anterior-posterior abdominal depth. It was determined by comparing the estimate to measured anterior-posterior abdominal depth (measured at the time of the x-ray examination). Results are expressed as a percentage deviation; a low % deviation is more accurate, a high % deviation less accurate.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: percentage agreement (est/measured)
Arm/Group | Patient Cohort
Number analyzed (Participants) | 20
percentage agreement (est/measured) | 5.8 (4.6)

ADVERSE EVENTS:
Time Frame: 1 day
Description: There was no harm possible as a result of this trial. Therefore, all-cause mortality, serious and other [not including serious] adverse events were not monitored or assessed.
Arm/Group | Patient Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03341546/Prot_SAP_000.pdf